CLINICAL TRIAL: NCT04046276
Title: Neuroprotective, Motor and Cognitive Impact of a Long-standing Aerobic Training Program in Parkinson's Disease. A Multicenter Comparison of the Effects of Two Aerobic Programs of Graded Intensities and a Conventional Physical Therapy Program Prolonged for 9 Months on Nigrostriatal, Motor and Cognitive Functions.
Brief Title: Intensity of Aerobic Training and Neuroprotection in Parkinson's Disease
Acronym: AEROPROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P140926; 2015-A01345-44 (Other: IDRCB)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Aerobic Exercises; High Intensity Training; Neuroprotection
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-blind randomized study, three parallel groups (n= 7 or 8 per group and per center, over 3 centers):
  * Group 1 "Conventional Physical Therapy", CPT
  * Group 2 "Medium Intensity Aerobic program", MIA (50% VO2 max);
  * Group 3 "High Intensity Aerobic program", HIA (70% VO2 max); HIA and MIA groups are experimental groups and CPT group is the control group. Each group will attend 3 weekly 45-minute sessions at the hospital for 9 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: * Study participants will be unaware of the hypothesis.
  * All investigator assessors, clinical, cardiological, biomechanical or through SPECT [123I] beta-CIT striatal uptake measurements, will be unaware of the participant group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physical Therapy (Placebo Comparator): Three sessions a week of hospital-based conventional physical therapy, all in presence and with the guidance of a registered physical therapist, for nine months
  Interventions: Other: Conventional Physical Therapy
- Medium Intensity Aerobic exercise (50% VO2 max) (Sham Comparator): Three sessions a week of hospital-based Medium Intensity Aerobic exercise (50% VO2 max); on a stationary bicycle, all in presence and with the guidance of a physical education teacher, for nine months
  Interventions: Behavioral: Medium Intensity Aerobic program
- High Intensity Aerobic exercise (Experimental): Three sessions a week of hospital-based High Intensity Aerobic exercise (70% VO2 max) on a stationary bicycle, all in presence and with the guidance of a physical education teacher, for nine months
  Interventions: Behavioral: High Intensity Aerobic program

INTERVENTIONS:
Behavioral: High Intensity Aerobic program — Three sessions a week of hospital-based exercise on a stationary bicycle, all in presence and with the guidance of a physical education teacher, for nine months
  Arms: High Intensity Aerobic exercise
Other: Conventional Physical Therapy — Three sessions a week of hospital-based exercise on a stationary bicycle, all in presence and with the guidance of a physical education teacher, for nine months
  Arms: Conventional Physical Therapy
Behavioral: Medium Intensity Aerobic program — Three sessions a week of hospital-based exercise on a stationary bicycle, all in presence and with the guidance of a physical education teacher, for nine months
  Arms: Medium Intensity Aerobic exercise (50% VO2 max)

SUMMARY:
In phenotypic animal models of Parkinson's Disease (PD), chronic physical exercise has produced nigrostriatal neuroprotection and symptom improvement, provided training was of high-intensity and prolonged duration (>3 months in rodent models). Conventional physical therapy in Parkinson's disease (PD) has traditionally avoided fatigue and high intensity workouts. Yet, in PD controlled studies have shown that: (i) an acute aerobic stress produces endogenous dopamine immediately after the exercise and (ii) short term (a few weeks) high intensity aerobic training enhances D2 striatal receptor density and cortical excitability and clinically improves walking, upper limb and executive functions; (iii) long-term (six months) high intensity aerobic treadmill training is associated with less deterioration of subjective UPDRS III score compared to a waiting list. Long-term high intensity aerobic training has not been compared to low or medium intensity training in PD patients for its objective motor, cognitive and putative neuroprotective effects.

DETAILED DESCRIPTION:
A short description, 5000 characters Intro: In phenotypic animal models of Parkinson's Disease (PD), chronic physical exercise has produced nigrostriatal neuroprotection and symptom improvement, provided training was of high-intensity and prolonged duration (>3 months in rodent models). Conventional physical therapy in Parkinson's disease (PD) has traditionally avoided fatigue and high intensity workouts. Yet, in PD controlled studies have shown that: (i) an acute aerobic stress produces endogenous dopamine immediately after the exercise and (ii) short term (a few weeks) high intensity aerobic training enhances D2 striatal receptor density and cortical excitability and clinically improves walking, upper limb and executive functions; (iii) long-term (six months) high intensity aerobic treadmill training is associated with less deterioration of subjective UPDRS III score compared to a waiting list. Long-term high intensity aerobic training has not been compared to low or medium intensity training in PD patients for its objective motor, cognitive and putative neuroprotective effects.

Hypothesis/Objective

Hypothesis High-intensity aerobic exercises practiced over 9 months will produce greater symptomatic motor and cognitive benefits and neuroprotective effects in PD patients, than low or medium intensity training.

Primary Objective To compare the motor effects of a 9-month conventional physical therapy program (light aerobic exercises), an aerobic program of medium intensity on stationary bicycle (50% maximal oxygen uptake, VO2 max), and an aerobic program of high intensity (70% VO2 max) in Parkinson's disease.

Secondary Objectives

* To evaluate aerobic capacities before and after the program.
* To evaluate cognitive functions, depression, quality of life before and after each program as well as 3 months following program termination and motor function 3 months following program termination.
* To explore potential neuroprotective effects of a 9-month aerobic program through specialized brain imaging (123I-Ioflupane SPECT) and a potential aerobic intensity-effect of such neuroprotection.

Primary outcome measure Change in MDS-UPDRS III Score (Movement Disorders Society - Unified Parkinson's Disease Rating Scale) in the " OFF " state between Day 1 and Month 9.

Secondary outcome measures OFF-state at Day 1, Month 9, Month 12

* Two-minute walking test from D1 to M9
* Modified 20-meter up-and-go test (AT20)
* 2-minute walk test (from M1 to M12)
* Global Mobility Task (GMT) scale (standing up off the floor)
* Upper limb performance in activities of daily living (Mount Sinai Parkinsonism Impairment Rating Scale, MSPIR)
* Static posturography
* Maximal aerobic capacity (VO2 max)
* Montreal Cognitive Assessment test (MoCA)
* Digit span task (forward and backward)
* Trail Making Test

ON-state at D1, M9, M12

* MDS-UPDRS III Score;
* Mean number of steps performed over the past three weeks (pedometry);
* Monthly incidence of falls in the past 3 months (questionnaire)
* Daily consumption of dopaminergic medications
* Quality of life (EQ-5D)
* Depression (GDS15)
* Dopaminergic striatal function by SPECT [123I] beta-CIT striatal uptake at D1, M12.

Method Design

Single-blind randomized study, 3 parallel groups (n= 7 or 8 per group and per center, over 3 centers):

* Group 1 " High Intensity Aerobic exercise ", HIA (70% VO2 max);
* Group 2 " Medium Intensity Aerobic exercise ", MIA (50% VO2 max);
* Group 3 " Conventional Physical Therapy ", CPT HIA and MIA groups are experimental groups and CPT group is the control group. Each group will attend 3 weekly 45-minute sessions at the hospital for 9 months.

Number of subjects needed: 69 Inclusion criteria Patients with diagnosis of PD according to the UKPDSBB criteria to distinguish idiopathic PD from atypical parkinsonism such as multi-system atrophy, progressive supra-nuclear paralysis or vascular parkinsonism; Previous MRI available, to further help distinguish idiopathic PD from atypical parkinsonism; Hoehn & Yahr Stage 1-3 in OFF state; Age > 18; Signed informed consent to participate in study.

Non-inclusion criteria Patients lacking motivation or ability to participate in training sessions for 9 months, in the investigator's opinion; contra-indications to high-intensity aerobic training in the cardiologist's opinion; contra-indications to perchlorate de potassium or to the use of 123I-FP-CIT; concurrent severe co-morbidities; cognitive deficit limiting participation to the program; Montreal Cognitive Assessment test (MoCA)<23; uninsured patient; participation in another ongoing interventional clinical trial (drug therapy, surgical treatment, another rehabilitation treatment, medical device); Pregnancy or current lactation, or no efficacious contraception during the 9 months of intervention.

Recruitment period: 1 year; Study duration: 26 months (24 patients recruited in 2 centers and 21 patients in the other 2 centers) Participation duration for each patient: 14 months Number of participating centers: 3

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the UKPDSBB criteria
* Previous MRI available, to further help distinguish idiopathic PD from atypical parkinsonism Hoehn & Yahr Stage 1-3 in OFF state
* Age > 18
* Signed informed consent to participate in study

Exclusion Criteria:

* Patients lacking motivation or ability to participate in training sessions for 9 months, in the investigator's opinion
* Contra-indications to high-intensity aerobic training in the cardiologist's opinion
* Contra-indications to perchlorate de potassium or to the use of 123I-FP-CIT
* Concurrent severe co-morbidities
* Cognitive deficit limiting participation to the program in the investigator's opinion
* Montreal Cognitive Assessment test (MoCA)<23
* Uninsured patient
* Participation in another ongoing interventional clinical trial (drug therapy, surgical treatment, another rehabilitation treatment, medical device)
* Pregnancy or current lactation, or no efficacious contraception during the 9 months of intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in MDS-UPDRS III Score (Movement Disorders Society - Unified Parkinson's Disease Rating Scale) in the " OFF " state between Day 1 and Month 9. | at day 1 and 9 Months
  The MDS-UPDRS III Score is a subjective assessment of motor symptoms based on the addition of ordinal 1-4 scores.

SECONDARY OUTCOMES:
Two-minute walking test at maximal speed | at day 1, 9 Months and 12 Months
Modified 20-meter up-and-go test (AT20) | at day 1, 9 Months and 12 Months
Global Mobility Task (GMT) | at day 1, 9 Months and 12 Months
  time required to stand up off the floor
Upper limb performance in activities of daily living (Mount Sinai Parkinsonism Impairment Rating Scale, MSPIR) | at day 1, 9 Months and 12 Months
  three unimanual tasks on each side and six bimanual everyday living tasks all times
Maximal aerobic capacity (VO2 max) | at day 1, 9 Months and 12 Months
Montreal Cognitive Assessment test (MoCA) | at day 1, 9 Months and 12 Months
Digit span task (forward and backward) | at day 1, 9 Months and 12 Months
Trail Making Test | at day 1, 9 Months and 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel GRACIES, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP)
Locations (3):
- France (3):
  - Henri Mondor Hospital, Créteil
  - Sébastopol hospital, Reims
  - Rangueil hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886